CLINICAL TRIAL: NCT07266272
Title: Influence of Extracorporeal Shockwave Therapy in Patients of Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mohamed Faramawy Shible El.deeb, Assistant lecturer of physical therapy for orthopedics and sport injuries, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Shockwave in neck pain
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Neck Pain Musculoskeletal; Neck Pain; Extracorporeal Shock Wave Therapy; Mechanical Neck Pain; Cervical Pain, Posterior; Pain Threshold
Keywords: Neck pain; Cervical joint position sense; Cervical range of motion; Pressure pain threshold; Extracorporeal shock wave therapy; Chronic mechanical neck pain
MeSH Terms: conditions — Neck Pain | interventions — Extracorporeal Shockwave Therapy; Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Statistician and outcome assessor who is also an investigator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group, standardized physiotherapy group receiving (Stretch, strength, Postural correction) (Other): The control group recieve conventional program without additional shockwave
  Interventions: Other: Exercise
- Intervention group received Extracorporeal shockwave therapy + Standardized physiotherapy as control (Experimental): Group B
  Interventions: Device: Extracorporeal Shockwave therapy; Other: Exercise

INTERVENTIONS:
Device: Extracorporeal Shockwave therapy — Radial, pneumatic extracorporeal shockwave therapy: The ESWT was applied using the following treatment parameters: 2,000 pulses, intensity of 1 to 1.2 bars, and 10 Hz frequency
  Other Names: ESWT
  Arms: Intervention group received Extracorporeal shockwave therapy + Standardized physiotherapy as control
Other: Exercise — Stretch + isometrics + postural correction
  Other Names: Strength _ Activation_ stretch_ postural correction

SUMMARY:
Purpose:

The study aimed to determine whether adding extracorporeal shockwave therapy (ESWT) to a standardized physiotherapy program provides additional benefits for patients with chronic mechanical neck pain. Specifically, it examined effects on pain intensity, pressure pain threshold (PPT), neck disability index (NDI), cervical active range of motion (AROM), and joint position sense (JPS).

DETAILED DESCRIPTION:
Study Summary Summary of the Study: Influence of Extracorporeal Shockwave Therapy in Patients with Mechanical Neck Pain

Purpose:

The study aimed to determine whether adding extracorporeal shockwave therapy (ESWT) to a standardized physiotherapy program provides additional benefits for patients with chronic mechanical neck pain. Specifically, it examined effects on pain intensity, pressure pain threshold (PPT), neck disability index (NDI), cervical active range of motion (AROM), and joint position sense (JPS).

Key Details:

* Study Design: Double-blinded, pretest-posttest controlled clinical trial.
* Participants: 52 patients aged 18-29 with chronic mechanical neck pain for over 3 months.
* Groups:

  * Group A: Standardized physiotherapy only (stretching, isometric exercises, posture training).
  * Group B: ESWT + standardized physiotherapy.
* Duration: 4 weeks, 2 sessions/week (1 ESWT + 1 physiotherapy in Group B).
* Assessments: NPRS for pain, pressure algometer for PPT, Arabic NDI, goniometer for AROM & JPS.
* Results:

  * Adding ESWT significantly improved PPT, left cervical rotation AROM, cervical extension JPS, and right cervical rotation JPS.
  * No significant differences between groups in other measures.
* Conclusion: ESWT combined with physiotherapy may enhance pain threshold, AROM in rotation, and proprioception compared to physiotherapy alone.

Sources of Strength in the Study:

1. Double-blind design reduces bias.
2. Randomized allocation with adequate sample size determined by power analysis.
3. Use of validated measurement tools (NPRS, NDI Arabic version, Wagner algometer, standard goniometer).
4. Clearly defined inclusion/exclusion criteria ensuring sample homogeneity.
5. Use of standardized physiotherapy protocol enhances reproducibility.

ELIGIBILITY:
Inclusion Criteria:

1. The patients (both males and females) with chronic non-specific neck pain for more than three months.
2. The patient's age is between 18 and 29 years old.
3. The patient has at least one taut band at the upper fibers of the trapezius as described in assessment procedures.
4. patient's numeric pain rating scale (NPRS) was 3 to 8 out of 10

Exclusion Criteria:

1. Were treated for neck or shoulder pain during the last three months.
2. Had a neck or shoulder operation during the last two years.
3. Had any structural pathology of the cervical spine, such as disk prolapse, spinal stenosis, or cervical spondylosis.
4. Had a traumatic history, instability, and spasmodic torticollis.
5. Had cardiovascular, respiratory, or allergic disease or neck osteoarthritis.
6. Had homeostatic disorders.
7. Fibromyalgia, shoulder diseases (tendonitis, bursitis, capsulitis).
8. Inflammatory rheumatic diseases.
9. Severe psychiatric illness and other diseases that restrict physical loading, and pregnancy (Salo et al., 2010).
10. Patients with vertebrobasilar insufficiency and vertigo.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold (PPT) | 4 weeks
  The minimum amount of pressure applied to body tissue that a person perceives as pain, rather than just pressure, is measured by an algometer. Another definition is the point at which a sensation changes from pressure to pain. measured by an algometer. A higher score is better, and a lower score is worse.

SECONDARY OUTCOMES:
Active cervical range of motion | 4 weeks
  Active cervical range of motion in 6 directions: flexion, extension, sidebending in both directions, and rotation in both directions. The higher score is better, and the lower score is worse.
Joint position sense | 4 weeks
  Joint position sense is measured by joint position error via the head repositioning test. The head repositioning test is the ability of the individual to detect the predetermined position again using the neck's sense of position and movement in 6 directions. The lower score is better, and the higher score is worse. The lowest score is zero.
Neck Pain | 4 weeks
  Pain is an unpleasant sensation measured by numeric pain rating score (NPRS) The highest score is 10, and the lowest score is zero. Ten is maximum pain, and zero is no pain. The higher score is worse, and the lower score is better.
Neck disability index (NDI) | 4 weeks
  The index displays the level of neck disability (questionnaire). The higher score is worse, and the lower score is better. Percentage score: The highest score is 100%, and the lowest score is 0%. Raw score: the lowest score is 0, and the highest score is 50.

CONTACTS AND LOCATIONS:
Locations (1):
- 12, Shibīn al Kawm, Menofya, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Akamatsu FE, Ayres BR, Saleh SO, Hojaij F, Andrade M, Hsing WT, Jacomo AL. Trigger points: an anatomical substratum. Biomed Res Int. 2015;2015:623287. doi: 10.1155/2015/623287. Epub 2015 Feb 24. PMID 25811029
- [Result] Abbott JH, Schmitt J. Minimum important differences for the patient-specific functional scale, 4 region-specific outcome measures, and the numeric pain rating scale. J Orthop Sports Phys Ther. 2014 Aug;44(8):560-4. doi: 10.2519/jospt.2014.5248. Epub 2014 May 14. PMID 24828475
- [Result] Abadiyan F, Hadadnezhad M, Khosrokiani Z, Letafatkar A, Akhshik H. Adding a smartphone app to global postural re-education to improve neck pain, posture, quality of life, and endurance in people with nonspecific neck pain: a randomized controlled trial. Trials. 2021 Apr 12;22(1):274. doi: 10.1186/s13063-021-05214-8. PMID 33845880
- [Result] Romeo P, Lavanga V, Pagani D, Sansone V. Extracorporeal shock wave therapy in musculoskeletal disorders: a review. Med Princ Pract. 2014;23(1):7-13. doi: 10.1159/000355472. Epub 2013 Nov 5. PMID 24217134
- [Result] Rahbar M, Samandarian M, Salekzamani Y, Khamnian Z, Dolatkhah N. Effectiveness of extracorporeal shock wave therapy versus standard care in the treatment of neck and upper back myofascial pain: a single blinded randomised clinical trial. Clin Rehabil. 2021 Jan;35(1):102-113. doi: 10.1177/0269215520947074. Epub 2020 Jul 30. PMID 32731757

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Shockwave in patients of neck pain protocol (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/72/NCT07266272/Prot_SAP_ICF_000.pdf